CLINICAL TRIAL: NCT02683473
Title: Measurement of Energy Metabolism in Infants: BabyEE Pilot
Brief Title: Measurement of Energy Metabolism in Infants
Acronym: BabyEE Pilot
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Leanne Redman, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 2015-061; P30DK072476-10 (NIH)
Record Dates: First submitted 2016-01-14; First posted 2016-02-17 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Infant Development; Infant Overnutrition
MeSH Terms: conditions — Infant Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants: Infants aged 1-3 months

SUMMARY:
The purpose of this study is to measure energy expenditure during the first 3 months of life in infants.

DETAILED DESCRIPTION:
This study intends to establish the feasibility of undertaking comprehensive metabolic phenotyping in infants. The overarching aim is to complete a prospective assessment of energy expenditure in the new infant metabolic chamber approximately one week apart to determine the accuracy and precision of infant protocols related to energy metabolism (sleeping metabolic rate, resting metabolic rate, diet-induced thermogenesis) and physical activity. This cross-sectional study will answer the following questions:

1. What is the test re-test reliability of measuring energy expenditure (sleeping metabolic rate, resting metabolic rate, diet-induced thermogenesis) in an infant under the same conditions, 5-7 days apart?
2. What is the reliability of 24h energy expenditure estimated by the infant metabolic chamber in comparison to a 7-day doubly labeled water study?
3. How do energy expenditure measurements in infants need to be adjusted to account for variability in infant size and body composition?

ELIGIBILITY:
Inclusion Criteria:

* Healthy, full-term infant
* Aged 1 month (28 days) to 3 months (12 weeks, 6 days) at the first visit
* Exclusively fed breast milk and/or infant formula
* Willing to accept doubly-labeled water

Exclusion Criteria:

* Unable to complete 3 clinic visits within about 14 days at Pennington Biomedical Research Center
* Born preterm (< 37 weeks gestation)
* Congenital abnormality or disability
* Gastric reflux
* Acute illness within 7 days of the study (fever, diarrhea)
* Use of medications to treat a chronic condition (does not include use of vitamin supplements or PRN medication for flatulence or reflux such as Pepcid)

Ages: 1 Month to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Full-term infants aged 1 to 3 months who are exclusively fed breast milk and/or infant formula will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-03-16 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Energy Expenditure by infant metabolic chamber | Approximately 1 week
  Energy expenditure by infant metabolic chamber measured twice about 1 week apart for test re-test reliability in infants aged 1-3 months.
Energy expenditure by doubly labeled water | Approximately 1 week
  Energy expenditure by doubly labeled water measured over 7 days in infants aged 1-3 months

SECONDARY OUTCOMES:
Percent body fat | Approximately 1 week
  Percent body fat by PEA POD measured twice about 1 week apart for test re-test reliability in infants aged 1-3 months.
Physical activity counts | Approximately 1 week
  Physical activity counts by Actigraph accelerometer measured over 7 days in infants aged 1-3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Redman, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No